CLINICAL TRIAL: NCT01605903
Title: Postoperative Ibuprofen and the Risk of Bleeding After Tonsillectomy With or Without Adenoidectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Hartnick, M.D., Associate Professor, Department of Otology and Laryngology; Chief, Division of Pediatric Otolaryngology; Director, Pediatric Airway, Voice and Swallowing Center, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-054H
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Tonsillectomy; Adenoidectomy
Keywords: Tonsillectomy; adenoidectomy; bleeding; bleeding rates; Tonsillectomy with and without adenoidectomy
MeSH Terms: conditions — Hemorrhage | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with Ibuprofen (Experimental): Children in the experimental group will receive grape-flavored ibuprofen 100mg/5 mL. Ibuprofen will be dispensed at 10mg/kg (max dose 600 mg) will be dispensed Q6 hours x 9 days.
  Interventions: Drug: Ibuprofen
- Treatment with Acetaminophen (Active Comparator): Children in the active comparator group will receive grape flavored acetaminophen 160 mg/5 ml. Acetaminophen will be dispensed at 15 mg/kg (max dose 650/mg) Q6 hours x 9 days.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Children in the ibuprofen group will be receive grape-flavored ibuprofen 100mg/5 mL. During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
  Other Names: Advil, Motrin
  Arms: Treatment with Ibuprofen
Drug: Acetaminophen — During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
  Other Names: Tylenol
  Arms: Treatment with Acetaminophen

SUMMARY:
Tonsillectomy (the surgical removal of the tonsils) is a commonly performed surgery in children. One risk of tonsillectomy is postoperative bleeding, and this can be more dangerous in children because their blood volume is lower than adults. Ibuprofen, a nonsteroidal anti-inflammatory medication (NSAID), is an effective pain medication. Recent guidelines, published by the American Academy of Otolaryngology, advocated use of ibuprofen after tonsillectomy. However, NSAIDs are associated with altered platelet function and a theoretical increased risk of bleeding after surgery. The investigators would like to explore the effect that ibuprofen has on postoperative bleeding, as well as validate previous studies demonstrating it is an effective pain medication after tonsillectomy.

DETAILED DESCRIPTION:
Tonsillectomy with and without adenoidectomy is one of the most commonly performed surgical procedures in the pediatric population. The incidence of adenotonsillectomy has increased over the past four decades (1). This is mainly due to increased awareness of the potential adverse consequences that pediatric sleep disordered breathing (SDB) may have on development and long-term pulmonary and cardiovascular health. SDB has surpassed recurrent tonsillitis as the most common indication for adenotonsillectomy in children (2-5). Over the past decade, according to the CDC's National Health Statistic Report on ambulatory surgery performed in the US, annual rates of tonsillectomy performed with and without adenoidectomy in children aged 15 and younger increased from 287,000 to 530,000 (6, 7). Adenotonsillectomy is the second most common procedure performed on children under the age of 15. Although generally considered a safe procedure, adenotonsillectomy has significant morbidity and potential for complications, particularly in the pediatric population. Complications include postoperative hemorrhage, dehydration, pain, anesthetic complications and airway risks, aspiration, and post-obstructive pulmonary edema (8). In young children, the risk of adenotonsillectomy is more critical due to smaller airways and respiratory reserve, as well as smaller blood volume (5).

Postoperative bleeding can be categorized as a primary event, occurring < 24 hours after surgery, or a secondary event, occurring >24 hours after tonsillectomy. Additionally, events can be further described by the interventions taken, such as emergency room visits, admission for observation, or return to the operating room to achieve hemostasis. Postoperative bleeding rates, including both primary and secondary events, range from 3.3-20%, with a mean of 4.5% (9). Thus, annually, tens of thousands of children experience exposure to potentially life-threatening postoperative hemorrhage, often requiring readmission, anesthetic exposure, and operative control of hemorrhage.

Postoperative pain contributes significantly to post-tonsillectomy morbidity. While narcotics are effective in controlling postoperative pain, they are often contraindicated, particularly in children with sleep disordered breathing, because of their potentially adverse side effects on respiration and the central nervous system (10). Nonsteroidal anti-inflammatories (NSAIDS), which block prostaglandin-induced inflammation and edema, are an attractive therapeutic option because they do not result in respiratory and central nervous system depression, and therefore may reduce the risk of postoperative respiratory depression, nausea and vomiting, excessive sedation and urinary retention. NSAIDS have been shown to be effective analgesics after tonsillectomy (11,12). However, because their mechanism of action may also interfere with platelet aggregation and increase bleeding time, their use is balanced with concern about an increased risk of postoperative hemorrhage. Aspirin, which irreversibly inhibits cyclooxygenase, affects coagulation and bleeding for up to 10 days, has been associated with an increased bleed rate after tonsillectomy (13). However, non-aspirin NSAIDs demonstrate a reversible inhibition of COX-1 and COX-2, and therefore do not have the same severe, prolonged effects on bleeding (14). Ibuprofen, a derivative of propionic acid, is widely used for musculoskeletal pain, but the study of its use for post-tonsillectomy analgesia is limited.

In 2011, The American Academy of Otolaryngology published Clinical Practice Guidelines outlining evidence-based selection and perioperative management strategies for tonsillectomy in children. As part of a recommendation that clinicians educate caregivers about the importance of postoperative pain management, Baugh et al advocated the use of ibuprofen postoperatively, stating, "ibuprofen can be used safely for pain control after surgery" (15), citing a 2005 Cochrane Review of NSAIDs and post-tonsillectomy bleeding in support of this guideline (16). The Cochrane Review recently added additional studies to their analysis and results remained similar. The most recent Cochrane Review, published in 2010, evaluated 15 randomized trials comparing NSAIDs with other analgesics or placebo, and determined that NSAID use did not significantly alter the number of perioperative bleeding episodes, both requiring and not requiring surgical intervention; this review did not distinguish between primary and secondary bleeding events (17). Because post-tonsillectomy hemorrhage is an uncommon event, a large number of participants is required to provide an adequate number of events to give a significant result, therefore the large sample size of >1000 children in the Cochrane Review is admirable. However, sample sizes were not adequate to compare the risk of bleeding with each individual NSAID. Additionally, NSAIDs were given in both oral and parenteral forms, as well as preoperatively, intraoperatively and postoperatively, and the duration of postoperative analgesic use differed between studies. The surgical technique used was not uniform between studies as well. It is our feeling that because of these limitations, the data is not sufficient to broadly implement the Academy's recommendation that ibuprofen can be safely used for post-tonsillectomy analgesia without more carefully controlled, prospective study.

Although there are many studies in the literature evaluating NSAID use after tonsillectomy, there are few randomized-prospective trials evaluating the use of ibuprofen, and few trials are powered to adequately assess the risk of postoperative hemorrhage. Designing and executing a study to specifically evaluate ibuprofen after pediatric tonsillectomy and rates of post-operative hemorrhage requiring return to the operating room for control is important to the pediatric otolaryngology community, particularly given the American Academy of Otolaryngology's recent clinical guidelines. The results of such a definitive study would possibly affect the tens of thousands of children at risk for post-tonsillectomy hemorrhage every year. It would affect our own standards of care as well as national and international norms.

Preliminary Studies:

At the Massachusetts Eye and Ear Infirmary there is no precedent for administering ibuprofen to children after tonsillectomy with or without adenoidectomy. Despite American Academy of Otolaryngology support for the use of ibuprofen in the postoperative setting, pediatric otolaryngologists at our institution are still hesitant to administer ibuprofen postoperatively without additional study of its use.

Within the Department of Pediatric Otolaryngology at the Massachusetts Eye and Ear Infirmary there is a precedent for successful completion of randomized, controlled trials involving adenotonsillectomy (19, 20). With principal investigators dedicated to clinical research, as well as research nurses and coordinators at our disposal, a prospective, controlled clinical trial of ibuprofen use after tonsillectomy can be implemented. Additionally, the Massachusetts Eye and Ear Infirmary calculates annual post-tonsillectomy hemorrhage rates, including percentage of patients returning to the emergency room for evaluation for possible post-operative bleeding, as well as the percentage of patients returning to the operating room for control of bleeding. Thus, there is a precedent for collecting data on postoperative bleeding events, as well as a controlled bleed rate to which prospective study hemorrhage rates can be compared.

The goal of our study is to determine if postoperative ibuprofen affects the rate of post-tonsillectomy hemorrhage using a non-inferiority trial design, which is intended to show that the effect of ibuprofen is no worse than acetaminophen, which will serve as our control. This differs from an equivalence trial, which aims to demonstrate that the experimental and control group do not differ more than a specified amount. The equivalence margin set for non-inferiority trials is often smaller than the treatment difference for which a placebo-controlled trial is powered, requiring a larger sample size. This will address two issues we have with the current literature evaluating NSAID use after tonsillectomy: inadequate sample size, and unrealistic treatment differences, including up to a 20% difference in bleed rates, required to detect a significant difference between NSAID and control groups. Because our trial will be designed to test non-inferiority, the null hypothesis will assume inferiority: the rate of hemorrhage requiring operative intervention in patients treated with postoperative ibuprofen after tonsillectomy will be increased compared to the rate in patients given acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 2-18 undergoing tonsillectomy with or without adenoidectomy by electrocautery alone for sleep disordered breathing or infectious tonsillitis will be included.
* Patients with complex medical conditions and craniofacial abnormalities will be included.
* Informed consent and child assent will be required for enrollment

Exclusion Criteria:

* Patients with a known personal or family history of a bleeding disorder will be excluded.
* Patients with a history of asthma, kidney or liver problems will also be excluded.
* Patients with tonsillectomy or adenoidectomy performed using a cold knife technique, microdebrider, coblation or plasma knife.
* Patients on NSAIDs for other medical conditions, or those who have taken NSAIDs within 1 week of surgery will be excluded.
* Patients with allergy to aspirin or other NSAIDs, acetaminophen, Red Dye #40 or Red Dye #33 will also be excluded.
* Pregnancy testing using urine β-subunit of hCG gonadotropin (beta-HCG) will be performed on all children > 13 years of age, or those younger than 13 who are menstruating; this is the testing protocol used at the Children's Hospital of Boston. Patients found to be pregnant will be excluded from participation.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 741 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (5):
- United States (5):
  - nited States Naval Medical Center, San Diego, San Diego, California
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Brook Army Medical Center, San Antonio, Texas
  - nited States Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Madigan Army Hospital, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erickson BK, Larson DR, St Sauver JL, Meverden RA, Orvidas LJ. Changes in incidence and indications of tonsillectomy and adenotonsillectomy, 1970-2005. Otolaryngol Head Neck Surg. 2009 Jun;140(6):894-901. doi: 10.1016/j.otohns.2009.01.044. PMID 19467411
- [Background] Bluestone CD. Current indications for tonsillectomy and adenoidectomy. Ann Otol Rhinol Laryngol Suppl. 1992 Jan;155:58-64. doi: 10.1177/00034894921010s112. PMID 1728903
- [Background] Tom LW, DeDio RM, Cohen DE, Wetmore RF, Handler SD, Potsic WP. Is outpatient tonsillectomy appropriate for young children? Laryngoscope. 1992 Mar;102(3):277-80. doi: 10.1288/00005537-199203000-00009. PMID 1545656
- [Background] Ross AT, Kazahaya K, Tom LW. Revisiting outpatient tonsillectomy in young children. Otolaryngol Head Neck Surg. 2003 Mar;128(3):326-31. doi: 10.1067/mhn.2003.60. PMID 12646834
- [Background] Randall DA, Hoffer ME. Complications of tonsillectomy and adenoidectomy. Otolaryngol Head Neck Surg. 1998 Jan;118(1):61-8. doi: 10.1016/S0194-5998(98)70376-6. PMID 9450830
- [Background] Blakley BW. Post-tonsillectomy bleeding: how much is too much? Otolaryngol Head Neck Surg. 2009 Mar;140(3):288-90. doi: 10.1016/j.otohns.2008.12.005. PMID 19248930
- [Background] Husband AD, Davis A. Pain after tonsillectomy. Clin Otolaryngol Allied Sci. 1996 Apr;21(2):99-101. doi: 10.1111/j.1365-2273.1996.tb01310.x. No abstract available. PMID 8735391
- [Background] Harley EH, Dattolo RA. Ibuprofen for tonsillectomy pain in children: efficacy and complications. Otolaryngol Head Neck Surg. 1998 Nov;119(5):492-6. doi: 10.1016/S0194-5998(98)70107-X. PMID 9807075
- [Background] St Charles CS, Matt BH, Hamilton MM, Katz BP. A comparison of ibuprofen versus acetaminophen with codeine in the young tonsillectomy patient. Otolaryngol Head Neck Surg. 1997 Jul;117(1):76-82. doi: 10.1016/S0194-59989770211-0. PMID 9230328
- [Background] REUTER SH, MONTGOMERY WW. ASPIRIN VS ACETAMINOPHEN AFTER TONSILLECTOMY. A COMPARATIVE DOUBLE-BLIND CLINICAL STUDY. Arch Otolaryngol. 1964 Aug;80:214-7. doi: 10.1001/archotol.1964.00750040220021. No abstract available. PMID 14160147
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Cardwell M, Siviter G, Smith A. Non-steroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003591. doi: 10.1002/14651858.CD003591.pub2. PMID 15846670
- [Background] Berkowitz RG, Zalzal GH. Tonsillectomy in children under 3 years of age. Arch Otolaryngol Head Neck Surg. 1990 Jun;116(6):685-6. doi: 10.1001/archotol.1990.01870060043006. PMID 2340121
- [Background] Schafer AI. Effects of nonsteroidal antiinflammatory drugs on platelet function and systemic hemostasis. J Clin Pharmacol. 1995 Mar;35(3):209-19. doi: 10.1002/j.1552-4604.1995.tb04050.x. PMID 7608308
- [Background] Lewis SR, Nicholson A, Cardwell ME, Siviter G, Smith AF. Nonsteroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2013 Jul 18;2013(7):CD003591. doi: 10.1002/14651858.CD003591.pub3. PMID 23881651
- [Background] Brigger MT, Cunningham MJ, Hartnick CJ. Dexamethasone administration and postoperative bleeding risk in children undergoing tonsillectomy. Arch Otolaryngol Head Neck Surg. 2010 Aug;136(8):766-72. doi: 10.1001/archoto.2010.133. PMID 20713751
- [Background] Lister MT, Cunningham MJ, Benjamin B, Williams M, Tirrell A, Schaumberg DA, Hartnick CJ. Microdebrider tonsillotomy vs electrosurgical tonsillectomy: a randomized, double-blind, paired control study of postoperative pain. Arch Otolaryngol Head Neck Surg. 2006 Jun;132(6):599-604. doi: 10.1001/archotol.132.6.599. PMID 16785404
- [Background] Collison PJ, Mettler B. Factors associated with post-tonsillectomy hemorrhage. Ear Nose Throat J. 2000 Aug;79(8):640-2, 644, 646 passim. PMID 10969475
- [Background] National Center for Health Statistics, Centers for Disease Control, Advance data 283: ambulatory surgery in the United States, 1994. National Center for Health Statistics. Available on the Web at www.cdc.gov/nchs.
- [Background] Cullen KA, Hall MJ, Golosinskiy A. Ambulatory surgery in the United States, 2006. Natl Health Stat Report. 2009 Jan 28;(11):1-25. PMID 19294964
- [Derived] Diercks GR, Comins J, Bennett K, Gallagher TQ, Brigger M, Boseley M, Gaudreau P, Rogers D, Setlur J, Keamy D, Cohen MS, Hartnick C. Comparison of Ibuprofen vs Acetaminophen and Severe Bleeding Risk After Pediatric Tonsillectomy: A Noninferiority Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2019 Jun 1;145(6):494-500. doi: 10.1001/jamaoto.2019.0269. PMID 30946442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 741 patients were enrolled between May 3, 2012 and January 20, 2017 at participating institutions (Massachusetts Eye and Ear Infirmary, Boston; Naval Medical Center San Diego, San Diego; Naval Medical Center Portsmouth, Portsmouth; and Madigan Army Medical Center, Tacoma) prior to surgery.
Pre-assignment Details: All enrolled subjects were randomized to a treatment group, however 53 (7.2%) patients did not receive the study medication , either because they dropped out prior to the first dose of study medication, the procedure was cancelled, alternative surgical technique was used, pharmacy error, or IV acetaminophen was administered.
Groups:
- Treatment With Ibuprofen: Children will be randomly assigned to receive either ibuprofen or acetaminophen prior to surgery.
  Ibuprofen: Children in the ibuprofen group will be receive grape-flavored ibuprofen 100mg/5 mL. During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
- Treatment With Acetaminophen: Children will be randomly assigned to receive either ibuprofen or acetaminophen prior to surgery.
  Acetaminophen: During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
Period: Overall Study
Arm/Group | Treatment With Ibuprofen | Treatment With Acetaminophen
Started | 345 | 343
Completed | 345 | 343
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Race and Ethnicity not collected
Groups:
- Treatment With Ibuprofen: Children will be randomly assigned to receive either ibuprofen or acetaminophen prior to surgery. Children in the ibuprofen group will be receive grape-flavored ibuprofen 100mg/5 mL. During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
  Ibuprofen: Children in the ibuprofen group will be receive grape-flavored ibuprofen 100mg/5 mL. During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
- Treatment With Acetaminophen: Children will be randomly assigned to either the treatment arm or active comparator prior to surgery. Children in the active comparator group (Acetaminophen) will receive grape flavored 160 mg/5 ml acetaminophen. Acetaminophen will be dispensed at 15 mg/kg (max dose 650/mg) Q6.
  Acetaminophen: During the postoperative period, ibuprofen 10mg/kg (max dose 600 mg) will be dispensed Q6.
- Total: Total of all reporting groups
Arm/Group | Treatment With Ibuprofen | Treatment With Acetaminophen | Total
Number analyzed (Participants) | 345 | 343 | 688
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [4 to 8] | 5 [3 to 7] | 5 [4 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 154 | 322
  Male | 177 | 189 | 366
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Level 3 Postoperative Hemorrhage
Description: Postoperative hemorrhage is defined as any history of bleeding occurring within the 14 day postoperative period. Hemorrhage will be stratified into 3 levels of severity. Level 1: includes children with a history of postoperative bleeding evaluated and/or treated by a physician in the emergency room, inpatient unit or operating room; Level 2: children requiring inpatient admission for postoperative bleeding regardless of the need for operative intervention; Level 3: children requiring inpatient admission and return to the operating room for control of post-tonsillectomy hemorrhage.
Time Frame: Data about post-tonsillectomy bleeding will be obtained after the end of a 14-day postoperative period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ibuprofen | Treatment With Acetaminophen
Number analyzed (Participants) | 345 | 343
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 14-day postoperative follow-up period.
Arm/Group | Treatment With Ibuprofen | Treatment With Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/345 | 0/343
Serious Adverse Events (participants affected / at risk) | 0/345 | 0/343
Other Adverse Events (participants affected / at risk) | 0/345 | 0/343

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2012-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT01605903/SAP_000.pdf
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT01605903/Prot_001.pdf